CLINICAL TRIAL: NCT05340101
Title: Effect of Progressive Muscle Relaxation Exercise on Primary Dysmenorrhea Menstrual Symptoms and Quality of Life. Randomized Controlled Study
Brief Title: Effect of Progressive Muscle Relaxation Exercise on Primary Dysmenorrhea Menstrual Symptoms and Quality of Life.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sidika Pelit Aksu, Research asistant (RN), Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 77082166
Record Dates: First submitted 2022-03-30; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Primary Dysmenorrhea; Quality of Life
Keywords: Dysmenorrhea; Quality of Life; Menstrual Symptoms; nursing students
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): This group will practiced progressive muscle relaxation exercise
  Interventions: Behavioral: ROGRESSIVE MUSCLE RELAXATION EXERCISE
- control group (No Intervention): This group will not practiced progressive muscle relaxation exercise

INTERVENTIONS:
Behavioral: ROGRESSIVE MUSCLE RELAXATION EXERCISE — In the application, "Relaxation Exercises CD Audio Recordings" prepared by the Turkish Psychological Association were used. In the the second part of 30 minutes were explained with the sound of the PKGE stream and verbal instructions. Audio recordings in the second part were used in this study. In line with the PCGE sound recordings, each muscle group starting from the hands to the feet, and then the facial and whole body muscles were stretched for about 10 seconds. The exercise was applied by taking deep breaths while tensing each muscle group, and releasing this breath slowly during relaxation. The relaxation lasted 10-20 seconds before the next muscle group was stretched. In this way, the muscles groups in the hands, arms, neck, shoulders, chest, abdomen, hips, feet and fingers, face and whole body were voluntarily stretched and relaxed, respectively, and the students were relaxed.
  Arms: experimental group

SUMMARY:
In this study, it was aimed to evaluate the effect of progressive muscle relaxation exercise on dysmenorrhea, menstrual symptoms and quality of life in university students with common primary dysmenorrhea. The research is a single center, parallel group block randomized controlled experimental study. This study will be conducted in the Department of Nursing, Faculty of Health Sciences, of a state university in Turkey. The universe of the research will be Gazi University Faculty of Health Sciences, third year and last year nursing students (N: 451). In order to determine the sample size in the research, power analysis was performed using the G Power 3.1.0 program. For this purpose, the study results of Sis Çelik and Ejder Apay (2021), which were similar to our study, were taken as reference. According to the power analysis made by calculating the effect size; It was determined that the sample of the study should consist of a total of 42 people, 21 in each group, will be randomized.

The data of the research; Personal information form will be collected using Visual Analogue Scale (VAS), SF-12 Quality of Life Scale Short Form, Menstrual Symptom Scale, Dysmenorrhea Monitoring Form. The implementation of the research is planned between April 15, 2022 and August 15, 2022. Third and fourth year nursing students will be included in the study. First of all, it will be evaluated according to the sampling inclusion criteria using the pre-evaluation form. Women who meet the inclusion criteria will be informed about the purpose and importance of the research, and women who agree to participate in the study will be determined. Informed consent form will be signed by the women who accepted to participate in the study, Visual Analogue Scale, Menstrual Symptom Scale and SF 12 Short Form will be applied. Randomization will be done after obtaining consent and filling out the forms.

DETAILED DESCRIPTION:
Non-pharmacological methods include body therapies, mind-body based therapies, Chinese herbal medicine and vitamin mineral supplements. In particular, physical exercises, acupuncture, aromatherapy, Chinese herbal medicine and yoga are non-pharmacological methods frequently used in the management of dysmenorrhea. Progressive muscle relaxation exercise (PMRE), one of the mind-body based therapies, is frequently used in pain management, but there are limited studies on its effect on primary dysmenorrhea. Progressive muscle relaxation exercise focuses on recognizing muscle tension and then reducing this tension. Studies conducted in different populations have found that progressive muscle relaxation exercise reduces pain and improves quality of life.

There is insufficient evidence for the effect of progressive muscle relaxation exercises in the management of primary dysmenorrhea. Therefore, in this study, it was aimed to evaluate the effect of progressive muscle relaxation exercise on dysmenorrhea, menstrual symptoms and quality of life in university students with common primary dysmenorrhea.

METHOD Type of Research The research is a single center, parallel group block randomized controlled experimental study.

Location and Characteristics of the Research This study will be conducted in the Department of Nursing, Faculty of Health Sciences, of a state university in Turkey.

Population and Sample of the Research The universe of the research will be Gazi University Faculty of Health Sciences, third year and last year nursing students (N: 451). In order to determine the sample size in the research, power analysis was performed using the G Power 3.1.0 program. For this purpose, the study results of Sis Çelik and Ejder Apay (2021), which were similar to our study, were taken as reference. According to the power analysis made by calculating the effect size; It was determined that the sample of the study should consist of a total of 24 participants, 12 in the intervention group and 12 in the control group (α=0.05, 1-β =0.99, Effect size d= 1.9111974, tail(s)=two). Considering the drop out rate of the study as 36%, a total of 42 people, 21 in each group, will be randomized.

Inclusion criteria for the study;

* Having primary dysmenorrhea,
* Being Nulligravida,
* Having a history of regular menstrual cycles in the last six months (cycle duration 21-35 days),
* Not using hormonal contraceptives,
* A score of 5 or more on the visual analog scale (VAS).
* Not to have metabolic disease, cancer, heart disease and diabetes, diagnosed psychiatric disease, and not using antidepressant medication that would prevent him from performing PCGE.
* Not doing any other body-mind based practice
* Using a smartphone
* Not having any communication problems (mental, auditory, visual, etc.)
* To be willing to participate in the study. Exclusion criteria,
* Use of complementary therapies, anti-inflammatory therapy, antidepressants or anxiolytics during the study
* Occurrence of menstrual cycle irregularity
* Performing PKGE 3 times a week or less in a row Validity-Reliability Selection criteria have been determined to prevent selection bias. Inclusion criteria for the study; Having primary dysmonaea, being nulligravida, having a history of regular menstrual cycles in the last six months (cycle duration 21-35 days), not using hormonal contraceptives, having a score of 5 or more on the visual analog scale (VAS) Metabolic disease that will prevent performing PCI, Not having cancer, heart disease and diabetes, not having a diagnosed psychiatric disease and not using antidepressant drugs, not using anti-inflammatory drugs, not using any other body-mind based application, using a smart phone, having any communication problems (mental, auditory, visual, etc.) .) and volunteering to participate in the study. Block randomization will be used for randomization. Permutation series and assignment list to be used for group assignments will be created in computer environment (www.randomizer.org).

In this study on application bias, researcher and participant blinding will not be done. Because the researcher will make the application himself and placebo cannot be used in the intervention. Blinding will not be done in this study.

Pre-tests to prevent detection bias and randomization assignment of women will be done by an independent nurse.

The data obtained from the research aimed at preventing reporting bias will be coded as A and B by an independent researcher and transferred to the SPSS program. Analysis of the data will also be done by an independent statistician.

In order to prevent attrition bias, Intention to Treat Test will be used in case of decrease/reduction in the sample group or if post-tests are not filled.

Application Data Collection Tools The data of the research; Personal information form will be collected using Visual Analogue Scale (VAS), SF-12 Quality of Life Scale Short Form, Menstrual Symptom Scale, Dysmenorrhea Monitoring Form.

Personal Information Form:

The personal information form consists of 27 questions. It was prepared by researchers in line with literature information in order to identify students with primary and secondary dysmenorrhea (Ferries-Rowe et al., 2020; ACOG, 2018). In addition, the sociodemographic characteristics of the students and their methods of coping with dysmenorrhea, if any, were also questioned in the prepared form. Students who do not meet the eligibility criteria of the study will be excluded.

Visual Analog Scale (VAS): In the 10 cm Visual Analog Scale (VAS), "0" indicates no pain and "10" indicates the most severe level of pain. As the score on the scale increases, the severity of the pain increases.

Short Form of Quality of Life Scale SF-12 It was created as a short form of SF-36, which was developed by Ware et al. in 1995 to evaluate quality of life. It contains the same sub-dimensions as the SF-36. The Turkish validity and reliability study of the SF-12 scale was conducted by Soylu and Kütük (2021). The scale is used in the evaluation of physical (FIM-12) and mental health (MBI-12), which are the two main components of general health status. The scale includes physical functionality (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functionality (1 item), emotional role (2 items), and mental health. It consists of 8 sub-dimensions, including health (2 items) and 12 items. The higher the score obtained from the scale, the higher the quality of life. The Cronbach's alpha value of the FIM-12 sub-dimension of the scale was 0.73, and the Cronbach's alpha value of the MDS-12 sub-dimension was 0.72.

Menstruation Symptom Scale The Menstruation Symptom Scale (MSI) was developed by Chesney and Tasto in 1975 to assess menstrual pain and symptoms. Turkish validity and reliability study Güvenç et al. (2014) by It consists of 3 sub-dimensions including Negative Effects/Somatic Complaints, Pain Symptoms and Coping Methods. The scale has a 5-point likert structure. The scale score is calculated by calculating the MSÖ score, the total score average of the items in the scale. An increase in the mean score indicates an increase in the severity of menstrual symptoms. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions. An increase in the score indicates that the severity of the symptoms in that sub-dimension increases. The total Cronbach's alpha value of the scale was found to be 0.92. The Cronbach's alpha value for the sub-dimensions was 0.90 for "Negative Effects/Somatic Complaints", 0.81 for "Pain Symptoms" and 0.74 for "Coping Methods".

Dysmenorrhea Monitoring Form: This form was prepared by the authors in accordance with the literature (Coşkuner and Kömürcü, 2014; Çelik and Apay 2021). The form provides a prospective measurement of pain intensity. Students in the experimental and control groups will be asked to record their initial (first three days of the first cycle) pain severity level on the VAS form. Progressive relaxation exercises will be used for two menstrual cycles in the experimental group. The students in the experimental group will be asked to record on the VAS the dysmenorrhea felt before and after PBGE in the first three days of the menstrual cycle. The control group would not receive any intervention for dysmenorrhea pain in the second and third cycles when they marked their pain level.

Progressive Muscle Relaxation Exercise Tracking Chart It was prepared by the researcher in order to facilitate the follow-up of female students' PCGE application status. At the top of the chart are the student's name-surname and the start date of the application. On the other hand, the table includes the application weeks and whether the PCG is applied or not. The duration of the schedule application will vary according to the length of the menstrual cycle. For each week, boxes have been created to mark the days of the week and whether the application has been made or not. In the first menstrual cycle after being included in the study, no marking will be made on the chart. From the end of the first cycle, progressive muscle relaxation exercise should be performed 4 times a week for two menstrual cycles and recorded in the chart.

Analysis of Data The data will be stored in the computer environment using the Statistical Package for Social Sciences 20 (SPSS 20) statistical program. Kolmogorov-Smirnov test will be performed in order to determine the conformity of the scale scores to the normal distribution. Non-parametric tests (Mann-Whitney U test, Wilcoxon Test) will be used in statistical analysis since it was determined that the scores were not suitable for normal distribution. Mean and standard deviation will be used in the evaluation of quantitative variables, and frequency and percentage values will be used in the evaluation of qualitative variables. The p=0.05 value will be accepted as statistical significance in all statistical analyses. The effect size was determined by calculating Cohen's d (small-0.2, medium-0.5 and large effect-0.8). The Cronbach-α coefficient will be used to evaluate the reliability of the scales used in the study.

Ethical Dimension of Research Before the application, written permission from the institution where the research was conducted, approval from the Ethics Committee and written informed consent from the students will be obtained. After the implementation of the research is over, it will be planned to teach and practice progressive muscle relaxation exercises to the students in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study;

  * Having primary dysmenorrhea,
  * Being Nulligravida,
  * Having a history of regular menstrual cycles in the last six months (cycle duration 21-35 days),
  * Not using hormonal contraceptives,
  * A score of 5 or more on the visual analog scale (VAS).
  * Not to have metabolic disease, cancer, heart disease and diabetes, diagnosed psychiatric disease, and not using antidepressant medication that would prevent him from performing PCGE.
  * Not doing any other body-mind based practice
  * Using a smartphone
  * Not having any communication problems (mental, auditory, visual, etc.)
  * To be willing to participate in the study. Exclusion criteria,
  * Use of complementary therapies, anti-inflammatory therapy, antidepressants or anxiolytics during the study
  * Occurrence of menstrual cycle irregularity
  * Performing PKGE 3 times a week or less in a row

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
change difference primary dysmenorrhea of the groups | 8 weeks
  Visual Analog Scale
change difference between the menstrual symptom scale scores of the groups | 8 weeks
  menstrual symptom scale

CONTACTS AND LOCATIONS:
Overall Officials: Sıdıka PELİT AKSU, PhD, Principal Investigator — Gazi University
Locations (1):
- Sıdıka PELİT AKSU, Ankara, Turkey/Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No